CLINICAL TRIAL: NCT03487263
Title: A Phase 1b, Open-Label, Dose-Escalation, Safety and Pharmacokinetic Study of IC14 in Motor Neurone Disease
Brief Title: Dose-Escalation, Safety and Pharmacokinetic Study of IC14 in Motor Neurone Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Implicit Bioscience (Industry)
Collaborators: Royal Brisbane and Women's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALS01
Record Dates: First submitted 2018-03-09; First posted 2018-04-04 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Motor Neuron Disease; Amyotrophic Lateral Sclerosis
Keywords: motor neurone disease; amyotrophic lateral sclerosis; IC14 [anti-CD14 (cluster of differentiation 14) monoclonal antibody]; monoclonal antibody; anti-CD14
MeSH Terms: conditions — Motor Neuron Disease; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Open-label, dose-escalation, safety and pharmacokinetic
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IC14 dose level 1 (Experimental): For the initial 3 patients: intravenous IC14 at a dosage of 2 mg/kg on Study Day 1, then 1 mg/kg once daily on Study Days 3-5 for 4 total doses
  Interventions: Biological: IC14
- IC14 dose level 2 (Experimental): For the subsequent 7 patients: intravenous IC14 at a dosage of 4 mg/kg/day on Day 1, followed by IC14 2 mg/kg/day on Days 2-4
  Interventions: Biological: IC14

INTERVENTIONS:
Biological: IC14 — chimeric monoclonal antibody against human IC14
  Other Names: monoclonal antibody against CD14

SUMMARY:
Ten patients with motor neurone disease (MND, also known as amyotrophic lateral sclerosis or ALS) will be successively enrolled to one of two dose levels of IC14 (human chimeric monoclonal anti-CD14) intravenously for four doses. Patients must be within 3 years of MND diagnosis and have adequate respiratory function. Safety, tolerability, immunogenicity, and PK/PD will be measured. To evaluate feasibility of the endpoints, additional endpoints of ALSFRS-R, respiratory function tests, disease biomarkers and patient-reported outcomes will be measured.

DETAILED DESCRIPTION:
The objectives of this study are to determine:

* The safety, tolerability and immunogenicity of IC14 in patients with motor neurone disease (MND).
* The pharmacokinetics and pharmacodynamics of IC14 in patients with MND.
* The preliminary effect of IC14 on the Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R) in patients with MND.
* The preliminary effect of IC14 on forced vital capacity (FVC) and other clinical markers of disease severity in patients with MND.
* The preliminary effect of IC14 on patient-reported outcome measures.
* The preliminary effect of IC14 on disease biomarkers.

Ten patients with MND will be sequentially assigned to receive one of two dose regimens of IC14 in an unblinded manner:

* For the initial 3 patients: IC14 at a dosage of 2 mg/kg on Study Day 1, then 1 mg/kg once daily on Study Days 3-5 for 4 total doses.
* For the subsequent 7 patients: IC14 at a dosage of 4 mg/kg on Study Day 1, then 2 mg/kg once daily on Study Days 2-4 for 4 total doses.

Study participation will continue until 28 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

A patient must fulfill all of the following criteria to be eligible for enrollment:

1. Signed informed consent prior to initiation of any study-specific procedures.
2. Familial or sporadic motor neurone disease (MND) defined as clinically possible, probable, or definite by Awaji-Shima Consensus Recommendations.
3. First symptoms of MND within 3 years of informed consent.
4. Age between 18 and 75 years at time of informed consent.
5. Seated Forced Vital Capacity (FVC) ≥ 65% of predicted value.
6. Not taking riluzole or on a stable dose of riluzole for at least 4 weeks prior to screening visit.
7. Adequate bone marrow reserve, renal and liver function:

   * absolute neutrophil count ≥ 1500/µL
   * lymphocyte count < 48%
   * platelet count ≥ 150,000/µL
   * hemoglobin ≥ 11 g/dL
   * Estimated glomerular filtration rate (eGFR) >= 40 mL/min/1.73 m2
   * Alanine aminotransferase (ALT) and/or Aspartate aminotransferase (AST) ≤ 2x upper imit of normal (ULN), total bilirubin ≤ 1.5x ULN
   * serum albumin ≥ 2.8 g/dL
8. Females of childbearing potential should be using and committed to continue using one of the following acceptable birth control methods:

   * Sexual abstinence (inactivity) for 1 month prior to screening through study completion; or
   * Intrauterine device (IUD) in place for at least 3 months prior to study through study completion; or
   * Stable hormonal contraception for at least 3 months prior to study through study completion; or
   * Surgical sterilization (vasectomy) of male partner at least 6 months prior to study.
9. To be considered of non-childbearing potential, females should be surgically sterilized (bilateral tubal ligation, hysterectomy, or bilateral oophorectomy at least 2 months prior to study) or be post-menopausal and at least 3 years since last menses.
10. Males with female partners of childbearing potential must use contraception through study completion.
11. Medically safe to have lumbar puncture to collect cerebrospinal fluid.
12. Able to give informed consent and able to comply with all study visits and all study procedures.

Exclusion Criteria:

A patient fulfilling any of the following criteria at screening is to be excluded from enrollment in the study:

1. Dependence on mechanical ventilation, defined as being unable to lay supine without it, unable to sleep without it, or continuous daytime use; presence of tracheostomy at screening; or presence of diaphragm pacing system at screening.
2. Treatment with a drug or device within the last 30 days that has not received regulatory approval.
3. Treatment within 12 months with immunomodulator or immunosuppressant agent (including but not limited to cyclophosphamide, cyclosporine, interferon-α, interferon-β-1a, rituximab, alemtuzumab, azathioprine, etanercept, infliximab, adalimumab, certolizumab, golimumab, anakinra, rilonacept, secukinumab, tocilizumab, mycophenolate mofetil, methotrexate, haematopoietic stem cell transplantation).
4. Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other opportunistic infections or major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks.
5. History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies.
6. Presence of any of the following clinical conditions:

   * Bleeding diathesis or receipt of anticoagulants within 7 days (or any other clinical condition that would, in the opinion of the investigator, place the patient at increased risk during lumbar puncture).
   * History of one or more of the following: cardiac insufficiency (New York Heart Association [NYHA] III/IV), uncontrolled cardiac arrhythmias, unstable ischemic heart disease, or uncontrolled hypertension (systolic blood pressure > 170 mmHg or diastolic blood pressure > 110 mmHg).
   * History of venous thromboembolic disease within 12 months, myocardial infarction, or cerebrovascular accident.
   * Unstable pulmonary, renal, hepatic, endocrine or hematologic disease.
   * Autoimmune disease, mixed connective tissue disease, scleroderma, polymyositis, or significant systemic involvement secondary to rheumatoid arthritis.
   * Evidence of active malignant disease, malignancies diagnosed within the previous 5 years, or breast cancer diagnosed within the previous 5 years (except skin cancers other than melanoma).
   * Human immunodeficiency virus infection or other immunodeficiency illness.
   * Unstable psychiatric illness defined as psychosis or untreated major depression within 90 days.
   * Drug abuse or alcoholism within the past 12 months.
   * Significant neuromuscular disease other than MND.
   * Other ongoing disease that may cause neuropathy, such as toxin exposure, dietary deficiency, uncontrolled diabetes, hyperthyroidism, cancer, systemic lupus erythematosus or other connective diseases, infection with HIV, hepatitis B virus (HBV), or hepatitis C (HCV), Lyme disease, multiple myeloma, Waldenström's macroglobulinemia, amyloid, and hereditary neuropathy.
7. Pregnancy or breastfeeding.
8. Deprivation of freedom by administrative or court order.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety, tolerability) | one month
  Number of participants with treatment-emergent adverse events (safety, tolerability) classified by MedDRA

SECONDARY OUTCOMES:
Treatment-related change in ALSFRS-R functional scale | one month
  Treatment-related change in Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R) [0 (worst) to 48 (best)]
Respiratory function | one month
  Treatment-related change in percent normal Forced Vital Capacity [0% (worst) to 100% (best)]
Muscle function | one month
  Treatment-related change in percent normal Sniff Nasal Pressure [0% (worst) to 100% (best)]
Quality of life measured by ALSSQOL | one month
  Treatment-related change in Amyotrophic Lateral Sclerosis Specific Quality of Life - Revised (ALSSQOL-R) [0 (worst) to 460 (best)]
Patient-reported outcome | one month
  Treatment-related change Edinburgh Cognitive and Behavioural Assessment Score (ECAS) [0 (worst) to 136 (best)]
Maximum Plasma Concentration (Cmax) | one month
  Maximum serum IC14 concentration (micrograms per milliliter)
Area Under the Curve (AUC) | one month
  Area Under the Curve for serum IC14 (microgram x hr/mL)
Monocyte CD14 Receptor Occupancy | one month
  Treatment-related change in percent monocyte CD14 receptor occupancy as a pharmacodynamic marker
Urinary p75 neurotrophin receptor (biomarker) | one month
  Treatment-related change in urinary concentration of urinary p75 neurotrophin receptor (NTR) (nanograms per milligram creatinine)
Neurofilament (biomarker) | one month
  Treatment-related change in concentration of neurofilament (picograms per milliliter)
Anti-drug antibodies | one month
  Development of human anti-monoclonal antibodies following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Henderson, MBBS, Principal Investigator — Royal Brisbane and Women's Hospital
Locations (1):
- Royal Brisbane and Women's Hospital, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henderson RD, Agosti JM, McCombe PA, Thorpe K, Heggie S, Heshmat S, Appleby MW, Ziegelaar BW, Crowe DT, Redlich GL. Phase 1b dose-escalation, safety, and pharmacokinetic study of IC14, a monoclonal antibody against CD14, for the treatment of amyotrophic lateral sclerosis. Medicine (Baltimore). 2021 Oct 22;100(42):e27421. doi: 10.1097/MD.0000000000027421. PMID 34678870